CLINICAL TRIAL: NCT02029742
Title: Hydroxyurea Adherence for Personal Best in Sickle Cell Treatment: HABIT
Acronym: HABIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Nancy Green, Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ7350; R21NR013745 (NIH)
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Medication adherence; Hydroxyurea; Community health worker intervention; Sickle Cell Treatment
MeSH Terms: conditions — Anemia, Sickle Cell; Medication Adherence | interventions — Community Health Workers; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Community Health Worker Intervention (Experimental): Community Health Workers will have scheduled interactions with subjects and will customize text messaging jointly with each youth and parent and initiate text message reminders to both parent and youth for months 4-6.
  Interventions: Behavioral: Community Health Worker (CHW)
- Education (Active Comparator): Those randomized to the Education group will continue usual care, and will be provided with educational materials about sickle cell disease and hydroxyurea use for children.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Community Health Worker (CHW) — CHWs will have scheduled interactions with subjects at home, by telephone or at Community League of the Heights (CLOTH), our partner community-based organization (CBO). CHWs will customize text messaging jointly with each youth and parent (Month 3) and text message reminders to both parent and youth will be implemented during Months 4-6. Subjects lacking a mobile phone or sufficient cell phone plan will be compensated to purchase or upgrade plans to accommodate texts.
  Arms: Community Health Worker Intervention
Behavioral: Education — Dyads randomized to the control group will continue usual clinic-based care, including monitoring and review of HbF levels, and similar frequency of clinic visits and access to sickle cell team staff. They will be provided with educational materials about sickle cell disease and hydroxyurea use for children.
  Arms: Education

SUMMARY:
The investigators propose that culturally aligned community-based interventions in our multi-ethnic sickle cell disease (SCD) population, augmented by task-focused communication technology, can improve self-managed adherence to hydroxyurea (HU) by decreasing barriers to use, supporting parent-youth partnerships for chronic disease self-management and reinforcing the behavior of daily medication use. Culturally aligned community health workers (CHW) are a well-established means to support chronic disease self-management by underserved families, in partnership with medical homes. CHWs can identify and address multiple barriers and reinforce developmentally appropriate self-management to help youth reach and maintain their best fetal hemoglobin (HbF) levels. However, this strategy alone may be insufficient to achieve daily HU adherence. The investigators therefore propose a feasibility trial to test the feasibility and acceptability of a structured intervention of CHW support to address existing barriers to improve HU use, augmented by daily cue-based parent and youth text message reminders, to efficiently extend CHW family support and reinforce family partnerships for self-management.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is an inherited disorder affecting the blood and causes anemia, painful sickle crises, organ damage, reduced quality of life and high health care use. Hydroxyurea (HU) is an oral medication that reduces disease symptoms and improves quality of life by increasing the amount of fetal hemoglobin in the blood. Despite the clinical promise of hydroxyurea, many children with SCD do make taking hydroxyurea a daily health habit. General barriers to medication adherence in underserved populations include lack of trust of medical staff, incomplete knowledge regarding benefits of hydroxyurea, and other factors that impede access to care such as transportation difficulties. Challenges specific to hydroxyurea use include understanding the importance of maximizing fetal hemoglobin levels and addressing concerns about hydroxyurea. Children and adolescents also require that a developmentally appropriate transition of self-management be established with their parents. Community-based health workers are a well established means to provide support for chronic disease management for underserved families and address multi-faceted barriers through culturally, behaviorally and developmentally aligned intervention. The investigators hypothesize that Community Health Workers support, augmented by daily task-focused communication technology, can improve self-managed adherence to hydroxyurea.

ELIGIBILITY:
Inclusion Criteria:

Youth:

1. Sickle type - homozygous sickle disease or sickle-beta thalassemia disease
2. Age 10 to 18 years
3. Currently prescribed hydroxyurea (HU) ≥18 months (for assessing historical hydroxyurea adherence and identify personal best)
4. ≥3 fetal hemoglobin assessments over past 12 months with pre-HbF ≥10% below historical personal best value
5. Youth has/uses cell phone with text message capability
6. Youth able to speak/read English or Spanish.
7. Youth willing to participate

Parent:

1. Parent/legal guardian meets all inclusion criteria
2. Parent/guardian speaks/reads English or Spanish
3. Parent/ legal guardian willing to participate
4. Family expected to reside in community for ≥ 1 years

Exclusion Criteria:

Youth:

1. A different sickle type
2. Youth < 10 years of age or ≥ 18 years of age
3. Youth not prescribed hydroxyurea, or on chronic transfusions
4. <3 fetal hemoglobin assessments over past 12 months
5. Sexually active female ≥11 not using reliable contraception (due to hydroxyurea teratogenic risk)
6. Pregnancy
7. Cognitive impairment (>1 level below expected grade)
8. Youth not residing with parent/legal guardian
9. Sibling of a youth enrolled in this study

Parent:

1. Parent/legal guardian is not the primary caregiver
2. Youth in foster care

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Effect size of the intervention on hydroxyurea (HU) adherence | 6 months
  In this feasibility study, feasibility will be assessed of our methods, the impact of the intervention on adherence to hydroxyurea, and the ability to retain subjects throughout the 6 month period. These data will be used to calculate the effect size of the intervention to estimate the sample needed for a larger trial.

SECONDARY OUTCOMES:
Effect size of the intervention on youth-parent communication about self-management responsibility | 6 months
  The investigators will estimate the effect size of the intervention on youth-parent communication about self-management responsibility by assessing quantitative changes in questionnaires administered to both parents and youth.
Effect size of the intervention on youth-parent communication about quality of life (QOL) | 6 months
  The investigators will estimate the effect size of the intervention on youth-parent communication about quality of life by assessing quantitative changes in in general pediatric and Sickle Cell disease Quality of Life questionnaires administered to both parents and youths.
Effect size of the intervention on youth-parent communication about resource use | 6 months
  The investigators will estimate the effect size of the intervention on youth-parent communication about resource use, such as urgent outpatient appointments, emergency room visits, hospitalizations, missed days from school and parent productivity by assessing quantitative changes in questionnaires administered to parents.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Green, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center - Albert Einstein College of Medicine, The Bronx, New York

REFERENCES:
- [Result] Smaldone A, Stockwell MS, Osborne JC, Cortes Y, Bekele E, Green NS. Adolescent and parent use of new technologies for health communication: a study in an urban latino community. J Public Health Res. 2015 Feb 19;4(1):376. doi: 10.4081/jphr.2015.376. eCollection 2015 Feb 20. PMID 25918691
- [Result] Bekele E, Thornburg CD, Brandow AM, Sharma M, Smaldone AM, Jin Z, Green NS. Do difficulties in swallowing medication impede the use of hydroxyurea in children? Pediatr Blood Cancer. 2014 Sep;61(9):1536-9. doi: 10.1002/pbc.25073. Epub 2014 Apr 17. PMID 24753149
- [Result] Green NS, Manwani D, Matos S, Hicks A, Soto L, Castillo Y, Ireland K, Stennett Y, Findley S, Jia H, Smaldone A. Randomized feasibility trial to improve hydroxyurea adherence in youth ages 10-18 years through community health workers: The HABIT study. Pediatr Blood Cancer. 2017 Dec;64(12):10.1002/pbc.26689. doi: 10.1002/pbc.26689. Epub 2017 Jun 23. PMID 28643377
- [Result] Osborne JC, Green NS, Smaldone AM. Quality of Life of Latino and Non-Latino Youth With Sickle Cell Disease as Reported by Parents and Youth. Hisp Health Care Int. 2020 Dec;18(4):224-231. doi: 10.1177/1540415320908525. Epub 2020 Mar 3. PMID 32124643
- [Result] Smaldone A, Findley S, Manwani D, Jia H, Green NS. HABIT, a Randomized Feasibility Trial to Increase Hydroxyurea Adherence, Suggests Improved Health-Related Quality of Life in Youths with Sickle Cell Disease. J Pediatr. 2018 Jun;197:177-185.e2. doi: 10.1016/j.jpeds.2018.01.054. Epub 2018 Mar 20. PMID 29571930
- [Result] Smaldone A, Manwani D, Green NS. Greater number of perceived barriers to hydroxyurea associated with poorer health-related quality of life in youth with sickle cell disease. Pediatr Blood Cancer. 2019 Jul;66(7):e27740. doi: 10.1002/pbc.27740. Epub 2019 Apr 2. PMID 30941907
- [Derived] Smaldone A, Findley S, Bakken S, Matiz LA, Rosenthal SL, Jia H, Matos S, Manwani D, Green NS. Study protocol for a randomized controlled trial to assess the feasibility of an open label intervention to improve hydroxyurea adherence in youth with sickle cell disease. Contemp Clin Trials. 2016 Jul;49:134-42. doi: 10.1016/j.cct.2016.06.004. Epub 2016 Jun 17. PMID 27327779